CLINICAL TRIAL: NCT02144220
Title: Remote Access to Care, Everywhere: Using Telemedicine to Deliver Patient-centered Care to Patients With Parkinson Disease
Brief Title: Remote Access to Care, Everywhere, for Parkinson Disease
Acronym: RACE-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Davis Phinney Foundation (Other)
Responsible Party: Principal Investigator, Ray Dorsey, Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RSRB-50627
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Parkinson Disease
Keywords: Telemedicine; Virtual care visit; Remote visit; Video-conferencing
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Virtual care visit (Experimental): One-time virtual care visit for Parkinson disease.
  Interventions: Other: Virtual care visit

INTERVENTIONS:
Other: Virtual care visit — Video-conferencing visit with a Parkinson disease specialist
  Other Names: Telemedicine visit; Virtual house call

SUMMARY:
The primary objective of this study is to evaluate the feasibility, efficacy and the value of providing care to individuals with Parkinson disease directly into their homes. The specific aims are:

1. To demonstrate the feasibility of conducting remote evaluations of patients with Parkinson disease nationally;
2. To measure the impact of remote care on each patient's ability to improve his or her quality of life (QoL) and better manage his or her Parkinson disease; and
3. To assess the long-term acceptability to patients in receiving ongoing care remotely via telemedicine.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 30
* Self reported diagnosis of idiopathic Parkinson disease
* Ability to converse in English
* Ability and willingness to provide informed consent and complete study requirements
* Access to a non-public computer or similar devices with broadband internet.
* Located in New York, Maryland, Delaware, California, or Florida at time of virtual visit (or veterans with Parkinson disease anywhere in the U.S.)

Exclusion Criteria:

* Any condition (e.g.prominent psychosis) that in the investigator's or coordinator's judgment would preclude participation.
* Concurrent enrollment in another telemedicine study.

Ages: 30 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2014-03; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Ray Dorsey, MD, MBA, Principal Investigator — University of Rochester
Locations (3):
- United States (3):
  - University of California San Francisco/San Francisco VA Medical Center, San Francisco, California
  - University of Florida, Gainesville, Florida
  - University of Rochester Medical Center, Rochester, New York

REFERENCES:
- [Background] Dorsey ER, Venkataraman V, Grana MJ, Bull MT, George BP, Boyd CM, Beck CA, Rajan B, Seidmann A, Biglan KM. Randomized controlled clinical trial of "virtual house calls" for Parkinson disease. JAMA Neurol. 2013 May;70(5):565-70. doi: 10.1001/jamaneurol.2013.123. PMID 23479138
- [Background] Venkataraman V, Donohue SJ, Biglan KM, Wicks P, Dorsey ER. Virtual visits for Parkinson disease: A case series. Neurol Clin Pract. 2014 Apr;4(2):146-152. doi: 10.1212/01.CPJ.0000437937.63347.5a. PMID 24790799
- [Background] Dorsey ER, Constantinescu R, Thompson JP, Biglan KM, Holloway RG, Kieburtz K, Marshall FJ, Ravina BM, Schifitto G, Siderowf A, Tanner CM. Projected number of people with Parkinson disease in the most populous nations, 2005 through 2030. Neurology. 2007 Jan 30;68(5):384-6. doi: 10.1212/01.wnl.0000247740.47667.03. Epub 2006 Nov 2. PMID 17082464
- [Background] Dorsey ER, George BP, Leff B, Willis AW. The coming crisis: obtaining care for the growing burden of neurodegenerative conditions. Neurology. 2013 May 21;80(21):1989-96. doi: 10.1212/WNL.0b013e318293e2ce. Epub 2013 Apr 24. PMID 23616157
- [Background] Willis AW, Schootman M, Evanoff BA, Perlmutter JS, Racette BA. Neurologist care in Parkinson disease: a utilization, outcomes, and survival study. Neurology. 2011 Aug 30;77(9):851-7. doi: 10.1212/WNL.0b013e31822c9123. Epub 2011 Aug 10. PMID 21832214
- [Background] Willis AW, Schootman M, Tran R, Kung N, Evanoff BA, Perlmutter JS, Racette BA. Neurologist-associated reduction in PD-related hospitalizations and health care expenditures. Neurology. 2012 Oct 23;79(17):1774-80. doi: 10.1212/WNL.0b013e3182703f92. Epub 2012 Oct 10. PMID 23054239
- [Background] The European Parkinson's Disease Association. The european parkinson's disease standards of care consensus statement. http://www.kompetenznetzparkinson.de/EPDA_Parkinson_s_Standard_nsus_Statement_Vol_I.pdf>2013.
- [Background] Biglan KM, Voss TS, Deuel LM, Miller D, Eason S, Fagnano M, George BP, Appler A, Polanowicz J, Viti L, Smith S, Joseph A, Dorsey ER. Telemedicine for the care of nursing home residents with Parkinson's disease. Mov Disord. 2009 May 15;24(7):1073-6. doi: 10.1002/mds.22498. PMID 19353687
- [Background] Dorsey ER, Deuel LM, Voss TS, Finnigan K, George BP, Eason S, Miller D, Reminick JI, Appler A, Polanowicz J, Viti L, Smith S, Joseph A, Biglan KM. Increasing access to specialty care: a pilot, randomized controlled trial of telemedicine for Parkinson's disease. Mov Disord. 2010 Aug 15;25(11):1652-9. doi: 10.1002/mds.23145. PMID 20533449
- [Derived] Korn RE, Wagle Shukla A, Katz M, Keenan HT, Goldenthal S, Auinger P, Zhu W, Dodge M, Rizer K, Achey MA, Byrd E, Barbano R, Richard I, Andrzejewski KL, Schwarz HB, Dorsey ER, Biglan KM, Kang G, Kanchana S, Rodriguez R, Tanner CM, Galifianakis NB. Virtual visits for Parkinson disease: A multicenter noncontrolled cohort. Neurol Clin Pract. 2017 Aug;7(4):283-295. doi: 10.1212/CPJ.0000000000000371. PMID 28840919

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was primarily online through mass email messaging from the Davis Phinney Foundation, internet listings on Fox Trial Finder, messages from PatientsLikeMe, Google AdWords in eligible states, and outreach to support groups.
Pre-assignment Details: Individuals indicated their interest in participating by either visiting the Davis Phinney Foundation's "funded research" web page where individuals completed an online screening survey or by contacting study coordinators by phone or email.
Period: Overall Study
Arm/Group | Virtual Care Visit
Started | 277
Completed | 258
Not Completed | 19
Not completed — technology incompatibility | 9
Not completed — Lack of Efficacy | 4
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Virtual Care Visit
Number analyzed (Participants) | 277
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (9.1)
Gender [Count of Participants; unit: Participants]
  Female | 138
  Male | 139
Region of Enrollment [Number; unit: participants]
  United States | 277

OUTCOME MEASURES:

1. Primary Outcome: Feasibility
Description: The percent of telemedicine visits completed as scheduled. (Goal >80%)
Time Frame: 6 months
Measure: Number; unit: percentage of visits
Arm/Group | Virtual Care Visit
Number analyzed (Participants) | 277
percentage of visits | 91

2. Primary Outcome: Change in Quality of Life as Measured by the PDQ-39 Assessment Tool
Description: The impact on Quality of life (QoL) as measured by the change in PDQ-39 score from baseline to 6 months. The PDQ-39 is a 39-item self-report questionnaire, which assesses Parkinson's disease-specific health related quality over the last month. 5-point ordinal scoring system: 0 = never, 1 = occasionally, 2 = sometimes, 3 = often, 4 = always. Each dimension total score range from 0 (never have difficulty) to 100 (always have difficulty). Lower scores reflect better quality of life.
Time Frame: Baseline and 6 months
Measure: Number (95% Confidence Interval); unit: units on a scale
Arm/Group | Virtual Care Visit
Number analyzed (Participants) | 258
units on a scale | 0.4 [-1.5 to 0.6]
Statistical Analysis 1: Comparison: Virtual Care Visit; Test type: Superiority or Other; p = 0.39, t-test, 2 sided

3. Secondary Outcome: Acceptability
Description: - The percent of patients participated who stated that they are interested in receiving ongoing care for their PD via telemedicine. (Goal >80%)
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Virtual Care Visit
Number analyzed (Participants) | 258
percentage of participants | 74

4. Secondary Outcome: Feasibility (Descriptive)
Description: Percentage of physician visits where the physician was were satisfied or very satisfied with the virtual visit overall.
Time Frame: 6 months
Measure: Number; unit: percentage of visits
Arm/Group | Virtual Care Visit
Number analyzed (Participants) | 258
percentage of visits | 94

5. Secondary Outcome: Percentage of Patients Who Felt That the Recommendations Improved Their Health
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Virtual Care Visit
Number analyzed (Participants) | 258
percentage of participants | 56

ADVERSE EVENTS:
Arm/Group | Virtual Care Visit
Serious Adverse Events (participants affected / at risk) | 0/277
Other Adverse Events (participants affected / at risk) | 0/277

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes